CLINICAL TRIAL: NCT03348397
Title: Contegra Versus Pulmonary Homograft for Right Ventricular Outflow Tract Reconstruction in Newborns : Fifteen Years' Experience
Brief Title: Contegra Versus Pulmonary Homograft for Right Ventricular Outflow Tract Reconstruction in Newborns
Status: Completed | Type: Observational
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2016/Cardio/RVOTtherapy
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Congenital Heart Defect; Right Ventricular Outflow Tract Reconstruction
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contegra patients
  Interventions: Procedure: right ventricular outflow tract reconstruction with contegra
- Pulmonary homograft patients
  Interventions: Procedure: right ventricular outflow tract reconstruction with pulmonary homograft

INTERVENTIONS:
Procedure: right ventricular outflow tract reconstruction with contegra — Contegra pulmonary valved conduit is an animal jugular vein that contains a valve with three leaflets that are similar to a human heart valve.
  Groups: Contegra patients
Procedure: right ventricular outflow tract reconstruction with pulmonary homograft — cryopreserved pulmonary homografts
  Groups: Pulmonary homograft patients

SUMMARY:
Pulmonary homografts are standard substitutes for right ventricular outflow tract reconstruction in congenital heart surgery. Unfortunately shortage and conduit failure secondary to early calcifications and shrinking are observed particularly for small sized conduits in younger patients. In neonates, Contegra® 12mm could be a valuable alternative, but conflicting evidence exists. This retrospective study compared the outcome of these two conduits in a newborn population.

ELIGIBILITY:
Inclusion Criteria:

neonatal patients who had a reconstruction of the right ventricular outflow tract with a pulmonary homograft or a Contegra between January 1992 and December 2014 at HUDERF

Exclusion Criteria:

NA

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who underwent a right ventricular outflow tract reconstruction between January 1992 and December 2014 at the Hôpital Universitaire des Enfants Reine Fabiola, Belgium
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Comparison of mid term course between pediatric right ventricular outflow tract recontruction with homograft and contegra | up to 195 months post right ventricular outflow tract recontruction

SECONDARY OUTCOMES:
Proportion of early conduit-related reintervention according to the Nakata index | up to 195 months post right ventricular outflow tract recontruction
Proportion of early conduit-related reintervention according to the congenital heart defect diagnosis | up to 195 months post right ventricular outflow tract recontruction
Proportion of early conduit-related reintervention in right ventricular outflow tract recontructed with contegra | up to 195 months post right ventricular outflow tract recontruction
Proportion of early conduit-related reintervention in right ventricular outflow tract recontructed with pulmonary homograft | up to 195 months post right ventricular outflow tract recontruction
Overal mortality in right ventricular outflow tract recontructed with contegra | up to 195 months post right ventricular outflow tract recontruction
Overal mortality in right ventricular outflow tract recontructed with pulmonary homograft | up to 195 months post right ventricular outflow tract recontruction
Residual pulmonary arterial hypertension rate in right ventricular outflow tract recontructed with contegra | up to 195 months post right ventricular outflow tract recontruction
Residual pulmonary arterial hypertension rate in right ventricular outflow tract recontructed with pulmonary homograft | up to 195 months post right ventricular outflow tract recontruction

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wauthy, MDPhD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falchetti A, Demanet H, Dessy H, Melot C, Pierrakos C, Wauthy P. Contegra versus pulmonary homograft for right ventricular outflow tract reconstruction in newborns. Cardiol Young. 2019 Apr;29(4):505-510. doi: 10.1017/S1047951119000143. Epub 2019 Apr 3. PMID 30942148